CLINICAL TRIAL: NCT00888004
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multiple Oral Dose Study to Assess the Efficacy and Tolerability of AFQ056 in Reducing L-dopa Induced Dyskinesias in Parkinson's Patients With Severe L-dopa Induced Dyskinesias
Brief Title: Efficacy and Safety of AFQ056 in Reducing L-dopa Induced Dyskinesias in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056A2206; 2008-006270-15
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease; L-dopa Induced Dyskinesia
Keywords: Parkinson's; L-dopa; dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Active (Experimental)
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056
  Arms: Active
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of administration of AFQ056 in combination with L-dopa, in reducing the number of L-dopa related dyskinesias in Parkinson's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease
* Patients with L-dopa induced dyskinesia for at least 3 months
* Patients with L-dopa treatment for at least 3 years, stable for 1 month minimum

Exclusion Criteria:

* History of severe allergy to food or drugs
* Very low or high body weight.
* Prior surgery for Parkinson's Disease
* Smokers Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Number and severity of Dyskinesias and the safety and tolerability of administering AFQ056 in combination with L-dopa | 20 days

SECONDARY OUTCOMES:
Safety and tolerability of administration of AFQ056 in combination with L-dopa | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Germany (5):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leun-Biskirchen
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Tübingen

REFERENCES:
- [Derived] Berg D, Godau J, Trenkwalder C, Eggert K, Csoti I, Storch A, Huber H, Morelli-Canelo M, Stamelou M, Ries V, Wolz M, Schneider C, Di Paolo T, Gasparini F, Hariry S, Vandemeulebroecke M, Abi-Saab W, Cooke K, Johns D, Gomez-Mancilla B. AFQ056 treatment of levodopa-induced dyskinesias: results of 2 randomized controlled trials. Mov Disord. 2011 Jun;26(7):1243-50. doi: 10.1002/mds.23616. Epub 2011 Apr 11. PMID 21484867